CLINICAL TRIAL: NCT04540965
Title: Double-Blind, Randomized, 2-Way Crossover Evaluation of the Impact of a Histamine-H2 Receptor Antagonist (H2RA) on the Pharmacokinetics of Telaglenastat Administered to Healthy Adult Subjects
Brief Title: Impact of a Histamine H2 Receptor Antagonist (H2RA) on the Pharmacokinetics (PK) of Telaglenastat in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: CX-839-015
Record Dates: First submitted 2020-08-19; First posted 2020-09-07 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Drug Interaction
MeSH Terms: interventions — CB-839; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Famotidine or Placebo for famotidine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Telaglenastat and Famotidine (Experimental): Famotidine
  Interventions: Drug: Telaglenastat; Drug: Famotidine
- Telaglenastat and Placebo for Famotidine (Placebo Comparator): Placebo for famotidine
  Interventions: Drug: Telaglenastat; Drug: Placebo for famotidine

INTERVENTIONS:
Drug: Telaglenastat — Glutaminase inhibitor
  Other Names: CB-839
Drug: Famotidine — Histamine-H2 Receptor Antagonist
  Other Names: Pepcid
  Arms: Telaglenastat and Famotidine
Drug: Placebo for famotidine — Placebo for Histamine-H2 Receptor Antagonist
  Arms: Telaglenastat and Placebo for Famotidine

SUMMARY:
This study is designed to formally evaluate the impact of famotidine, an H2R antagonist, on the pharmacokinetics of telaglenastat.

This study will be conducted in up to 22 healthy volunteers, who meet all of the inclusion criteria and none of the exclusion criteria. The study is double-blinded, randomized 2-way crossover in design.

Subjects will receive four 200 mg tablets of telaglenastat either in the presence or absence of 20 mg famotidine (H2R-antagonist) with a 4-day wash-out period in between each regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female, 18-55 years of age, inclusive, at screening.
2. Has not used nicotine-containing products (more than 5 cigarettes/equivalent per week) for at least 3 months prior the first dose and has negative urine cotinine tests at screening, Day 1 and Day 7.
3. Body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusively, at screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECGs, as deemed by the Principal Investigator (PI).
5. For a female of childbearing potential: either be sexually inactive (abstinent - ie, not sexually active with a male partner) for 14 days prior to the first dose and through 14 days following the last dose of any study drug(s) or be using one of the following acceptable birth control methods:

   1. Non-hormone releasing intrauterine device in place for at least 3 months prior to the first dose of any study drug with a physical barrier method (eg, condom, diaphragm) from the time of screening through the last dose of any study drug. A progesterone (progestin)-only contraceptive is allowable.
   2. A physical barrier method (eg, condom, diaphragm) for at least 14 days prior to the first dose of any study drug and until the last dose of any study drug.
6. In addition, female subjects of childbearing potential will be advised to remain sexually inactive or to keep the same birth control method until the last dose of any study drug.
7. Females of non-childbearing potential as defined below do not require contraception.

   Females of non-childbearing potential:
   1. must have undergone one of the following sterilization procedures at least 6 months prior to the first dose of any study drug:

      1. hysteroscopic sterilization;
      2. bilateral salpingectomy;

   <!-- -->

   1. Women with a tubal ligation less than one year prior to study start must agree to use a barrier method of birth control 3. non-surgical transcervical sterilization (eg, Essure®); 4. hysterectomy; 5. bilateral oophorectomy OR
   2. be postmenopausal with amenorrhea for at least 1 year prior to the first telaglenastat dose with follicle-stimulating hormone (FSH) serum levels > 30 IU/mL.
8. A non-vasectomized male subject must agree to use a physical barrier (eg, condom or diaphragm) or abstain from sexual intercourse with female partners during the study until the last dose of any study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to study start. A male who has been vasectomized less than 4 months prior to study start must follow the same restrictions as a non-vasectomized male).

   a) Female participants with a vasectomized male partner, or male participants with a female partner of non-childbearing potential do not require contraception.
9. If male, must agree not to donate sperm from dosing until the last dose of any study drug.
10. Alanine and aspartate aminotransferase and bilirubin levels ≤ the upper limit of normal or deemed not clinically significant by the Investigator.
11. Understands the study procedures in the informed consent form (ICF) and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or is expected to manifest significant emotional problems during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI.
3. History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to screening.
5. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or inactive ingredient(s).
6. History or presence of:

   1. liver disease, pancreatic insufficiency or intestinal malabsorption;
   2. neuropathy or muscle disorders;
   3. seizures;
   4. asthma; childhood asthma that has resolved and has not required medical treatment for at least 5 years prior to study start is permitted;
   5. fluid retention;
   6. cardiovascular disease, cardiac arrhythmias, hypertension, cardiovascular thrombotic events, myocardial infarction, or stroke;
   7. ulcer disease or gastrointestinal bleeding;
   8. renal papillary necrosis and other renal injury;
   9. exfoliative dermatitis, Stevens-Johnson syndrome, and toxic epidermal necrolysis.
7. Female subjects who are pregnant or lactating.
8. Positive urine drug or alcohol results at screening or check-in.
9. Positive urine cotinine at screening or check-in.
10. Positive results at screening for HIV types 1 and 2, HBsAg, or hepatitus C virus.
11. Seated blood pressure (taken after 5 minutes in a sitting position) is less than 90/40 mmHg or greater than 140/90 mmHg at screening and not as part of ECG.
12. Seated heart rate (taken after 5 minutes in a sitting position) is lower than 40 bpm or higher than 100 bpm at screening and not as part of ECG.
13. QTcF interval is > 460 msec (males) or > 480 msec (females) or deemed clinically abnormal by the PI at screening.
14. Estimated creatinine clearance < 90 mL/min calculated by the method of Cockcroft and Gault at screening.
15. Unable to refrain from or anticipates the use of:

    1. Proton pump inhibitors (PPIs), histamine H2 receptor antagonists (H2RAs), buffering agents (eg, Tums) or any other medication that may have an effect on gastric acid secretion beginning 14 days prior to the first dose of any study drug and throughout the study.
    2. Any non-prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dose of any study drug and throughout the study.
    3. Any prescription medications (including hormone replacement therapy and lithium) beginning 14 days prior to the first dose of any study drug and throughout the study.
16. Donation of blood or significant blood loss within 56 days prior to the first dose of any study drug.
17. Plasma donation within 14 days prior to the first dose of any study drug.
18. Presence of any medical history or condition that may limit gastric drug absorption (eg, prior gastric surgery, gastric banding, Whipple procedure)
19. Participation in another clinical trial within 28 days prior to the first dose of any study drug. The 28-day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Blood samples taken on Day 3 and Day 9 at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24 hours post administration of the telaglenastat
  To assess the effect of famotidine on the Cmax of telaglenastat in healthy adult subjects
Time to peak plasma concentration (Tmax) | Blood samples taken on Day 3 and Day 9 at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24 hours post administration of the telaglenastat
  To assess the effect of famotidine on the Tmax of telaglenastat in healthy adult subjects
Area under the concentration-time curve from time = 0 to the last determination (AUClast) | Blood samples taken on Day 3 and Day 9 at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24 hours post administration of the telaglenastat with and without famotidine.
  To assess the effect of famotidine on the time to maximum plasma concentration (Tmax) of telaglenastat in healthy adult subjects.
Area under the concentration-time curve from time = 0 to infinity (AUC0-inf) | Blood samples taken on Day 3 and Day 9 at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24 hours post administration of the telaglenastat with and without famotidine.
  To assess the effect of famotidine on the AUC0-inf of telaglenastat in healthy adult subjects
Half-life | Blood samples taken on Day 3 and Day 9 at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24 hours post administration of the telaglenastat with and without famotidine.
  To assess the effect of famotidine on the half-life of telaglenastat in healthy adult subjects
Elimination rate | Blood samples taken on Day 3 and Day 9 at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24 hours post administration of the telaglenastat with and without famotidine.
  To assess the effect of famotidine on the elimination rate of telaglenastat in healthy adult subjects

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Safety will be assessed throughout the study, starting from Day 3, prior to receiving the first dose of telaglenastat through to Day 11 when the subjects are released from the clinical site.
  Assessed by physician reports of any unfavorable and unintended sign, symptom, or disease (new or exacerbated) that is temporally associated with the use of the investigational products.
Incidence of changes in body temperature | Body temperature will be assessed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Body temperature is measured in degrees Celsius.
Incidence of changes in respiratory rate. | Respiratory rate will be assessed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Respiratory rate is measured in breaths per minute.
Incidence of changes in blood pressure | Blood pressure will be assessed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Blood pressure is measured in mmHg.
Incidence of changes in heart rate. | Heart rate will be assessed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Heart rate is measured in beats per minute.
Electrocardiograms (ECGs) | ECGs will be performed prior to and 4 hours after telaglenastat dosing on Days 3 and 10 and 24 hours after telaglenastat dosing on Days 4 and 11.
  Triplicate 12-lead ECGs including P Wave, QRS Complex, and QTcF determination
Hemoglobin assessments | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Hemoglobin will be measured in g/dL
Hematocrit assessments | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Hematocrit will be measured in %
Leukocyte count assessments | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Leukocyte count will be measured in 1000 cells/microliter
Red blood cell count assessments | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Red blood cell count will be measured in 1,000,000 cells/microliter
Platelet count assessments | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Platelet count.will be measured in 1000 cells/microliter
Serum urea | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Serum Urea will be measured in mg/dL
Serum bilirubin | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Serum Bilirubin will be measured in micromoles/L
Serum alkaline phosphatase | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Serum alkaline phosphatase will be measured in units/L
Serum Aspartate aminotransferase assessments | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Serum Aspartate aminotransferase will be measured in units/L
Serum aspartate aminotransferase | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Serum Alanine aminotransferase will be measured in units/L
Serum albumin | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Serum Albumin will be measured in g/dL
Serum sodium | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Serum Sodium will be measured in meq/L
Serum potassium | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Serum Potassium will be measured in meq/L
Serum chloride | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Serum Chloride will be measured in meq/L
Serum glucose | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Serum Glucose will be measured in mg/dL
Serum creatinine | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Serum Creatinine will be measured in mg/dL
Urine pH | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Urine pH will be measured in units
Urine Specific gravity | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Urine Specific gravity will be measured in g/mL
Urine Protein | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Urine Protein will be measured in mg/24 hr
Urine Glucose | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Urine Glucose will be measured in mg/dL
Urine Ketones | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Urine Ketones will be measured in mg/dL
Urine Bilirubin | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Urine Bilirubin will be measured in mg/dL
Urine Blood | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Urine Blood will be measured in RBC/high powered field
Urine Nitrite | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Urine Nitrite will be measured by dipstick
Urine Urobilinogen | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Urine Urobilinogen will be measured in Ehrlich units
Urine Leukocyte esterase. | Assessments will be performed prior to dosing with telaglenastat on Days 2 and 9 and 24 hours after dosing on Days 4 and 11.
  Urine Leukocyte esterase will be measured in units

CONTACTS AND LOCATIONS:
Overall Officials: Paul Griffin, Dr., Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network Brisbane Clinic (formerly Q-Pharm), Brisbane, Queensland, Australia